CLINICAL TRIAL: NCT04752124
Title: Effect of High Intensity Speed Based Treadmill Training on Balance, Walking Capacity, and Quality in People With Sub-acute Stroke.
Brief Title: Effects of High-intensity Aerobic Training on Balance, Walking Capacity, and Quality of Life in Patients With Sub-acute Stroke.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Ishtiaq Ahmed, Physiotherapist, Government College University Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 555
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Stroke
Keywords: Cerebrovascular accident; Aerobic exercise; High intensity interval training
MeSH Terms: conditions — Stroke | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT+CT (Active Comparator): HIIT combined with conventional rehabilitation.
  Interventions: Other: Exercise Therapy; Other: conventional therapy
- Conventional therapy (Placebo Comparator): Conventional rehabilitation will be provided to this group of patients.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: Exercise Therapy — High intensity speed based interval treadmill training
  Arms: HIIT+CT
Other: conventional therapy — conventional physical therapy

SUMMARY:
Stroke is one of the major cause of morbidity and mortality and the leading cause of disability in adults all around the world. Stroke survivors can suffer several neurological impairments and deficits which have an important impact on patient's quality of life and which increase the costs for health and social services. After stroke, impairments in ADLs and functional status, deterioration in health related quality of life can be seen.

The purpose of this study is to Determine the effect of high intensity speed based treadmill training on Balance, Walking capacity and quality of life in sub-acute stroke.

ELIGIBILITY:
Inclusion Criteria:

* age 40-80 years; first episode of stroke; >4 weeks of stroke onset; hemiparesis resulting from unilateral ischaemic stroke; Ashworth score of 0 or 1, indicating no spasticity or slight spasticity over the affected lower limb, respectively; mini-mental state examination score ≥23; ability to perform independent walking for at least five minutes with or without an assistive device (FAC=3). All patients will be determined to be in stable cardiovascular condition with a low although slightly greater risk for vigorous exercise than for apparently healthy persons (class B according to the American College of Sports Medicine [ACSM]).13

Exclusion Criteria:

* Participants will be excluded from the study if they had any of the following: (1) chronic cardiorespiratory or metabolic diseases; (2) severe osteoporosis; and (3) lesions pertaining to the brainstem or cerebellum; (4) having resting blood pressure above 160/100 mmHg even after taking medications; (5) cardiovascular comorbidity (aortic stenosis, depression of ST-segment, heart failure, arrhythmias, unstable angina, hypertrophic cardio-myopathy); (6) transient ischemic attack; (7) by-pass surgery in the recent three months; and (8) other musculoskeletal problems that prevented the participants from doing aerobic activity.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-07 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | 6 weeks of training
  To determine the endurance after stroke

SECONDARY OUTCOMES:
Berg Balance scale | 5 weeks
  It is used to measure the Balance and stability of patient. Total score of the scale is 56. A score of < 45 indicates individuals may be at greater risk of falling.
Stroke Impact scale | 5 weeks
  To measure the impairment and quality of life after stroke. The maximum score is 140.

CONTACTS AND LOCATIONS:
Locations (1):
- Bin Inam Rehabilitation Center., Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lau KW, Mak MK. Speed-dependent treadmill training is effective to improve gait and balance performance in patients with sub-acute stroke. J Rehabil Med. 2011 Jul;43(8):709-13. doi: 10.2340/16501977-0838. PMID 21698340